CLINICAL TRIAL: NCT04015193
Title: Follow-up of Single-port Thoracoscopic Sympathicotomy in Patients With Raynaud's Phenomenon
Brief Title: Follow-up of SPTS in Patients With Raynaud's Phenomenon
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, dr. DJ Mulder, Vascular internist, Principal investigator, University Medical Center Groningen
Other Study IDs: 201900110
Record Dates: First submitted 2019-04-01; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Raynaud Phenomenon
MeSH Terms: conditions — Raynaud Disease | interventions — Patient Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Full responders: Full responders: no signs or symptoms of Raynaud's phenomenon (RP) in Raynaud condition score, no RP during cooling-recovery experiment.
  Interventions: Procedure: Single-port thoracoscopic sympathicotomy (patient care)
- Partial responders: Partial responders: at least 25% reduction in Raynaud condition score and finger ischemia time during cooling and recovery.
  Interventions: Procedure: Single-port thoracoscopic sympathicotomy (patient care)
- Non-responders: Non-responders: no or less than 25% reduction in Raynaud condition score and/or finger ischemia time during cooling and recovery.
  Interventions: Procedure: Single-port thoracoscopic sympathicotomy (patient care)

INTERVENTIONS:
Procedure: Single-port thoracoscopic sympathicotomy (patient care) — Single-port thoracoscopic sympathicotomy will be performed as part of patient care, data will be collected of patients undergoing this procedure

SUMMARY:
Background: Raynaud's phenomenon is a vasospasm of the extremities, leading to extensive discomfort in daily life and potentially severe ischemia. Some patients are resistant to conventional vasodilatory drug treatment. In the University Medical Center Groningen, single-port thoracoscopic sympathicotomy (SPTS) was developed. This is a new minimally invasive endoscopic technique, extensively limiting surgical burden. In many hospitals in the Netherlands, this operation is sometimes performed on patients with Raynaud's phenomenon. However, the techniques used are more invasive than the SPTS technique. Furthermore, studies on sympathectomy and sympathicotomy in Raynaud's are limited and encompass obsolete more invasive techniques. Also, it is unclear which patients would benefit the most and for how long and in which percentage of patients treatment effects persist over time. In a recent study on the new SPTS technique, it was found that one month after the procedure, the Raynaud's attacks were substantially reduced and the hand perfusion increased on the operated side. Based on these short term effects and previously reported broad experience with this technique for other indications, it is possible to offer this option to a broader range of patients with Raynaud's as a reasonable and safe treatment option. However, whether the effects persist on the long-term needs to be established.

Main research question: The aim of the study is to assess the 5 year efficacy and outcome in patients with primary and secondary Raynaud's phenomenon in whom SPTS has been performed.

Design (including population, confounders/outcomes): Patients with Raynaud's, who will undergo SPTS in patient care setting, will be included. Data from the patient file will be collected, including vascular measurements to assess hand perfusion, a Raynaud diary (Raynaud condition score, duration and frequency of the attacks), quality of life questionnaires, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Raynaud's phenomenon of the hands
* Scheduled SPTS as treatment for RP
* Age ≥ 16 years

Exclusion Criteria:

• SPTS for other indications than RP

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Raynaud's phenomenon
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Mean finger ischemia time | 5 year
  Mean finger ischemia time of five fingers during cooling and recovery, as assessed by routine cooling and recovery photo-electric plethysmography (PPG) after 5 years of follow-up, in minutes

SECONDARY OUTCOMES:
Mean finger ischemia time | 2 year
  Mean finger ischemia time of five fingers during cooling and recovery, as assessed by routine cooling and recovery photo-electric plethysmography (PPG) after 2 years of follow-up, in minutes
Raynaud Condition Score | 1,2,3,4,5 years
  Mean Raynaud condition score (0-100) over a period 14 days
Number of attacks | 1,2,3,4,5 years
  Mean number of RP attacks per day over a period of 14 days
Duration of attacks | 1,2,3,4,5 years
  Mean duration of RP attacks per day over a period of 14 days in minutes
SF-36 | 1,2,3,4,5 years
  Health-related quality of life short form (SF)-36 score of 100-0
HAQ | 1,2,3,4,5 years
  (Dutch) health assessment questionnaire (HAQ) score of 0-3
Capillary density | 2 and 5 years
  Mean number of capillaries per finger of 8 fingers per 3mm
Number of dilated capillaries | 2 and 5 year
  Mean number of dilated capillaries per finger (apex width >20µm, <50µm) of 8 fingers per 3mm
Number of giant capillaries | 2 and 5 year
  Mean number of giant capillaries per finger (apex width >50µm) of 8 fingers per 3mm
Capillaroscopic pattern | 2 and 5 year
  Pattern of nailfold capillaries (normal, non-specific, early, active or late)
Pulse wave velocity brachial-radial | 2 and 5 years
  Pulse wave velocity in m/s of brachial-radial trajectory
Systolic blood pressure | 2 and 5 years
  Brachial systolic blood pressure in mmHg
Diastolic blood pressure | 2 and 5 years
  Brachial diastolic blood pressure in mmHg
Mean finger blood pressure | 2 and 5 years
  Mean finger blood pressure in mmHg of eight fingers
Pulse wave velocity brachial-ulnar | 2 and 5 years
  Pulse wave velocity in m/s of brachial-ulnar trajectory
Digital ulcers | 1,2,3,4,5 years
  Incidence of digital ulcers (yes/no)
Compensatory sweating | 1,2,3,4,5 years
  Compensatory sweating (yes/no)
Wound infection or other adverse events | 2 weeks, 1,2,3,4,5 years
  Occurrence of wound infection or other adverse events potentially related to SPTS

CONTACTS AND LOCATIONS:
Overall Officials: Douwe J Mulder, MD, PhD, Principal Investigator — University of Groninge, University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided